CLINICAL TRIAL: NCT02412345
Title: Extracorporeal Shockwave Therapy in the Treatment for Erectile Dysfunction in Male Renal Transplant Recipients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Kleiton Gabriel Ribeiro Yamaçake, MD, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 41528915.5.0000.0068; 964.653 (Other: number of the opinion of the committee of ethics and research)
Record Dates: First submitted 2015-03-15; First posted 2015-04-09 (Estimated); Last update posted 2018-05-02 (Actual); Status verified 2018-05

CONDITIONS: Erectile Dysfunction; Renal Transplant
Keywords: Erectile Dysfunction; Shockwave therapy; Renal Transplant; Male; Renal Transplant Recipients
MeSH Terms: conditions — Erectile Dysfunction | interventions — Extracorporeal Shockwave Therapy; Alprostadil

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Extracorporeal Shockwave therapy (Experimental): Extracorporeal shockwave therapy at the penis. 6 sessions.
  Interventions: Procedure: Extracorporeal shockwave therapy; Other: Penile ultrasound Doppler with intracavernosal injection application 20 mcg alprostadil
- Sham treatment (Sham Comparator): Extracorporal shockwave therapy with a placebo probe. 6 sessions
  Interventions: Procedure: Extracorporeal shockwave therapy - sham treatment; Other: Penile ultrasound Doppler with intracavernosal injection application 20 mcg alprostadil

INTERVENTIONS:
Procedure: Extracorporeal shockwave therapy
  Arms: Extracorporeal Shockwave therapy
Procedure: Extracorporeal shockwave therapy - sham treatment — A probe similar to the treatment group will be used. The noise and appearance is similar. The probe emits zero energy during each treatment. Local application generates noise and a feeling of popping at the application site which will also be experienced by patients in the placebo group being impossible for the patient to discern which treatment group belongs.
  Arms: Sham treatment
Other: Penile ultrasound Doppler with intracavernosal injection application 20 mcg alprostadil — Diagnostic test will be performed before treatment and after 3 to 4 months after therapy.

SUMMARY:
The primary objective of this study is to determine the impact of the shock wave application in renal transplant patients with diagnosis of erectile dysfunction. Secondary objectives are to assess the effects of therapy on quality of life and depression.

It is expected that with the study is defined the usefulness of the therapy and the dissemination of knowledge generated for change in clinical management in renal transplant patients with erectile dysfunction.

DETAILED DESCRIPTION:
The Renal Transplant Unit, performs about 230 kidney transplants per year and has a screening service for registration of candidates for renal transplantation, interviewing about 70 patients a month. Since the potential and likely benefits of extracorporeal shock wave therapy in these patients as well as the anticipation of mild side effects, there is no reason for refusal to participate in the study.

Patients who meet the inclusion criteria will be divided into 2 groups using a randomization table created by computer. Patients will be followed for 2 years.

The study procedure and monitoring will be performed on an outpatient basis.

Patients are divided into a group of extracorporeal shockwave (ESWT) treatment and placebo in a ratio of 1: 1 using a table of random numbers generated by computer.

The ESWT protocol is protocol-based suggested by Vardi et al. 6. Patients will undergo a 2 treatment sessions per week for 3 weeks.

The penis is pulled manually, and shock waves are applied throughout the penile shaft (except the glans) and the crura bilaterally. The duration of each ESWT session will be approximately 10 minutes and 2000 shocks will be applied per session with an intensity of energy of 1 mJ / mm 2. The volume of penile tissue exposed to shock waves at each site will be cilyndric (diameter: 18 mm, height 100 mm). No local or systemic analgesia is required during the procedure.

To placebo therapy will be used the same device. The effective probe will be replaced by a similar one that emits zero energy during each treatment. Local application generates noise and a feeling of popping at the application site which will also be experienced by patients in the placebo group being impossible for the patient to discern which treatment group belongs.

Penile ultrasound Doppler and drug erection will be performed before therapy and after treatment to evaluate the results.

The diameter of the cavernous arteries is measured before and after intracavernosal injection application 20 mcg alprostadil (Caverject ®). In addition, vascular disorders, or stenotic atheromatous lesions will be investigated. The systolic and diastolic velocities of the cavernous arteries are evaluated 5,10 and 15 minutes after drug injection.

After obtaining the patient signed informed consent , will be included in the study. Laboratory tests will be held at the Hospital Laboratory.

Studied variables

The following parameters will be studied during the initial evaluation and follow-up:

1. Clinical

   Quality of life questionnaire -WHO QOL (World Health Organization - Quality of Life) Sexual questionnaire IIEF (International Index of Erectile Function) Comorbidities such as hypertension, diabetes and cardiovascular disease Smoking
2. Laboratory

   Total testosterone, free testosterone, progesterone, albumin, SHBG, FSH, LH, prolactin, complete blood count, urea, creatinine, total cholesterol and fractions, triglycerides, T3, T4F and TSH.
3. Imaging tests

Ultrasound Doppler penile before and 3 months after treatment.

- Calculation sample

To define the sample size, the investigators must take into account: data variability (within each group) and the difference the investigators want to observe the parameters to be studied before and after treatment, beyond the level of significance and power of the test.

The investigators will assume that the data follow a normal distribution and will use the paired t-test methodology, considering that the same patients will be evaluated in both conditions.

The level of significance that work is 5%. Suitable power will be considered to be greater than 80%.

The investigators observe a difference to 5 points required amount of samples is very small, whereas only 3 patients t-test. for the non-parametric test we consider a sample of 4 patients.

ELIGIBILITY:
Inclusion Criteria:

* Male patients between 40 and 70 years
* Kidney transplant for at least 6 months
* Erectile dysfunction (ED) for at least 6 months.
* Patients with IIEF score <21
* Functioning kidney graft.

Exclusion Criteria:

* ED because of known endocrine disease (e.g., hypogonadism, hypothyroidism)
* ED due to drug treatment (androgen deprivation therapy, for example)
* ED due to neurological disease (spinal cord injury, for example)
* ED due to structural abnormality of the penis
* History of radical prostatectomy or other pelvic surgery
* History of pelvic irradiation
* penile implant
* coagulopathies or on anticoagulants

Ages: 40 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-01; Primary Completion 2018-05-01 (Actual); Study Completion 2018-05-01 (Actual)

PRIMARY OUTCOMES:
Changing in International Index of Erectile Function (IIEF-5) from baseline | 1 month, 3 months, 6 months, 1 year, 2 years
Changing in Erection Hardness score from baseline | 1 month, 3 months, 6 months, 1 year, 2 years
Changing in The World Health Organization Quality of Life (WHOQOL) from baseline | 1 month, 3 months, 6 months, 1 year, 2 years
Changing in Peak systolic velocity by Penile doppler ultrasonography | baseline ( previous to treatment) and 3 months after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Kleiton Gabriel Ribeiro Yamaçake, São Paulo, Brazil

REFERENCES:
- [Background] Vardi Y, Appel B, Jacob G, Massarwi O, Gruenwald I. Can low-intensity extracorporeal shockwave therapy improve erectile function? A 6-month follow-up pilot study in patients with organic erectile dysfunction. Eur Urol. 2010 Aug;58(2):243-8. doi: 10.1016/j.eururo.2010.04.004. Epub 2010 May 6. PMID 20451317
- [Background] Yee CH, Chan ES, Hou SS, Ng CF. Extracorporeal shockwave therapy in the treatment of erectile dysfunction: a prospective, randomized, double-blinded, placebo controlled study. Int J Urol. 2014 Oct;21(10):1041-5. doi: 10.1111/iju.12506. Epub 2014 Jun 17. PMID 24942563
- [Background] Liu J, Zhou F, Li GY, Wang L, Li HX, Bai GY, Guan RL, Xu YD, Gao ZZ, Tian WJ, Xin ZC. Evaluation of the effect of different doses of low energy shock wave therapy on the erectile function of streptozotocin (STZ)-induced diabetic rats. Int J Mol Sci. 2013 May 21;14(5):10661-73. doi: 10.3390/ijms140510661. PMID 23698784